CLINICAL TRIAL: NCT05062811
Title: The Relationship Between Blood Pressure and Myocardial Work in Patients With Different Levels of Blood Pressure
Brief Title: Effect of Blood Pressure on Myocardial Work in Patients With Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Professor, Chongqing Medical University
Other Study IDs: MW-China2021
Record Dates: First submitted 2021-09-14; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Hypertension; Heart Disease, Hypertensive
MeSH Terms: conditions — Hypertension; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertension is a serious threat to human health and a major global economic burden. Chronic hypertension can cause left ventricular remodeling and loss of function, eventually leading to heart failure. Exploring the early changes and mechanisms of left ventricular cardiac function caused by hypertension, and to identify individuals who may develop into serious heart injury, may play a positive role in the early prevention and control of heart failure caused by hypertension. Therefore, this study intend to use two dimensional speckle tracking technology, a non-invasive method to measure left ventricular pressure-strain loop to quantitatively reflect cardiac work index , to study different hypertension patients with normal left ventricular ejection fraction the change of the global and local cardiac work, and the influence of aterosclerosis in the patients to myocardial work, and explore their relationship with ventricular remodeling and abnormal diastolic function. To improve the understanding of the pathophysiology of hypertension, hypertensive heart disease and heart failure, and to provide scientific support for the early prevention and control of such diseases. Myocardial work analysis Echocardiography plays a central role in the evaluation of patients with cardiovascular disease. Echocardiography is widely available and allows characterization of the functional and structural of heart. Thus, assessment of left lentricular (LV) global longitudinal strain (LVGLS) and Myocardial work indexes has proven benefit for both diagnosis and risk in hypertension patients.

DETAILED DESCRIPTION:
Hypertension is a serious threat to human health and a major global economic burden.Chronic hypertension can cause left ventricular remodeling and loss of function, eventually leading to heart failure. Ventricular remodeling in hypertensive patients is an adaptive and decompensating response to persistent elevated blood pressure and increased myocardial work load. Exploring the early changes and mechanisms of left ventricular cardiac function caused by hypertension, and to identify individuals who may develop into serious heart injury, may play a positive role in the early prevention and control of heart failure caused by hypertension.Therefore, this study intend to use two dimensional speckle tracking technology, a non-invasive method to measure left ventricular pressure-strain loop to quantitatively reflect cardiac work index , to study different hypertension patients with normal left ventricular ejection fraction (including hypertension without heart damage performance with different degree of high blood pressure, hypertension with diastolic dysfunction , hypertension with left ventricular hypertrophy ) the change of the global and local cardiac work, and the influence of aterosclerosis in the patients to myocardial work, and explore their relationship with ventricular remodeling and abnormal diastolic function.To improve the understanding of the pathophysiology of hypertension, hypertensive heart disease and heart failure, and to provide scientific support for the early prevention and control of such diseases.Now days, Echocardiography plays a central role in the evaluation of patients with cardiovascular disease. Echocardiography is widely available and allows characterization of the functional and structural of heart. Thus, assessment of left lentricular (LV) global longitudinal strain (LVGLS) and Myocardial work indexes has proven benefit for both diagnosis and risk in hypertension patients. Myocardial work indexes have four indexes to evaluate different function of lentricular. However, there is still no research investigating the the relationship between blood pressure and Myocardial work indexes in patients with different levels of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1.patients of outpatient clinic 2.65≥Adult aged ≥18years old;

Exclusion Criteria:

The exclusion criteria were patients aged less than 18 or greater than 65 years, previous diagnosis of diabetes mellitus, coronary artery disease, valve heart disease, primary cardiomyopathies, arterial fibrillation, left ventricular ejection fraction<50% , inadequate echocardiographic imaging. The patients with disease leading low PP(≤30mmHg) were special examined and excluded, including pericardial disease, severe mitral stenosis, aortic stenosis, severe chronic heart failure, blood loss and shock etc. A total of 40 patients were exclude from the study according to the preset criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension patients evaluated by echocardiography in the Echocardiography Center of the First Affiliated Hospital of Chongqing Medical University from September 2021 to January 2022.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Global work index | On admission
  Global work index by non-invasive pressure-strain loops: a novel parameter to assess left ventricular performance in the early stages of heart failure with preserved or mid-range ejection fraction after acute myocardial infarction
Global constructed work | On admission
  Global constructive work represented the sum of positive work due to myocardial shortening during systole and negative work due to lengthening during isovolumic relaxation.
Global longitudinal strain | On admission
  The assessment of global longitudinal strain (GLS) from speckle-tracking analysis of 2-dimensional echocardiography has become a clinically feasible alternative to LVEF for the measurement of myocardial function.

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No